CLINICAL TRIAL: NCT02572492
Title: Phase II Study of Carfilzomib-cyclophosphamide-dexamethasone and High-dose Melphalan (HDT) Followed by Randomization Between Observation or Maintenance With Carfilzomib and Dexamethasone in Patients With Relapsed Multiple Myeloma After HDT
Brief Title: Study of Carfilzomib in Multiple Myeloma Relapsed After High-dose Melphalan With Autologous Stem Cell Support
Acronym: CARFI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henrik Gregersen (Other)
Collaborators: Nordic Myeloma Study Group (Other)
Responsible Party: Sponsor-Investigator, Henrik Gregersen, Consultant, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMSG#20/13; 2013-003789-15 (EudraCT Number)
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Recurrence; Carfilzomib; Salvage Therapy; Transplantation, Autologous
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Neoadjuvant Therapy; carfilzomib; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carfilzomib/dexamethasone maintenance (Experimental): Carfilzomib/dexamethasone maintenance after salvage HDT
  Interventions: Drug: Induction with CAR-CY-DEX and conditioning with carfilzomib and highdose melphalan; Drug: Carfilzomib/dexamethasone maintenance
- Observation without maintenance (Sham Comparator): Observation without maintenance after salvage HDT
  Interventions: Drug: Induction with CAR-CY-DEX and conditioning with carfilzomib and highdose melphalan; Drug: Observation without carfilzomib/dexamethasone maintenance

INTERVENTIONS:
Drug: Induction with CAR-CY-DEX and conditioning with carfilzomib and highdose melphalan — All patients entering the study receive four series of CAR-CY-DEX (Cycle 1 with iv carfilzomib 20 mg/sqm on days 1 and 2, and iv carfilzomib 36 mg/sqm on days 8, 9, 15 and 16. Cycle 2 - 4 with iv carfilzomib 36 mg/sqm on days 1, 2, 8, 9, 15 and 16. P.o. cyclophosphamide 300 mg/sqm on days 1, 8 and 15 and p.o. dexamethasone 20 mg on days 1, 2, 8, 9, 15 and 16 in each 28-days series)
  Subsequently all patients receive the conditioning regimen:
  Iv carfilzomib 27 mg/sqm on day -2 and -1 Iv melphalan 200 mg/sqm on day -2 > 2.0 m CD34+ stem cells/kg body weight on day 0
  Other Names: Kyprolis
Drug: Carfilzomib/dexamethasone maintenance — Maintenance therapy two months after salvage HDT with iv carfilzomib 27 mg/sqm every second week and p.o. dexamethasone 20 mg every second week. The maintenance dose of carfilzomib will be escalated to 56 mg/sqm after 4 weeks provided acceptable side effects.
  Other Names: Kyprolis
  Arms: Carfilzomib/dexamethasone maintenance
Drug: Observation without carfilzomib/dexamethasone maintenance — Observation without carfilzomib/dexamethasone maintenance
  Arms: Observation without maintenance

SUMMARY:
This study evaluates induction therapy with carfilzomib-cyclophosphamide-dexamethasone before salvage high-dose melphalan with autologous stem cell support (HDT) in multiple myeloma patients with relapse after HDT done at diagnosis. In addition, the study evaluates the effect of maintenance therapy after salvage HDT in multiple myeloma. After salvage HDT half of the patients receive maintenance therapy with carfilzomib/dexamethasone while the other half are observed without maintenance therapy.

DETAILED DESCRIPTION:
The survival in younger myeloma patients improved in the nineties with the introduction of high-dose melphalan with autologous stem cell support (HDT) and despite the emergence of novel therapies HDT remains a keystone in myeloma treatment. However, all patients will eventually experience relapse after HDT performed at diagnosis. Eligible patients with late relapse are considered for salvage HDT. The duration of response after salvage HDT is in most studies reported to be approximately half the length of the response after initial HDT. The choice of induction treatment before HDT might affect the outcome after the induction therapy as well as the outcome after the HDT. In other settings the novel proteasome inhibitor Carfilzomib has showed superiority to the first-in-class proteasome inhibitor bortezomib. In addition, carfilzomib has a favourable profile of side effects. Thus, the aim of this phase 2 study is to evaluate induction therapy with carfilzomib-cyclophosphamide-dexamethasone before salvage HDT. The primary end-point in this part of the study is comparison of time to progression after the initial HDT and time to progression after salvage HDT when four series of carfilzomib-cyclophosphamide-dexamethasone are used as induction therapy. In the study Carfilzomib is also included in the conditioning regimen with administration of Iv carfilzomib 27 mg/sqm on day -2 and -1. The standard conditioning regime consists of Iv melphalan 200 mg/sqm on day -2 and reinfusion of at least 2.0 x 10m CD34+ stem cells/kg body weight on day 0.

The purpose of maintenance therapy in multiple myeloma is to prolong the time to progression of disease. There are limited data on the impact of maintenance therapy after salvage HDT. Another important aim of the study is therefore to evaluate the effect of carfilzomib/dexamethasone given every other week compared to observation without maintenance therapy. This part of the study starts two months after HDT. The randomization is stratified according to relapse 1 - 2 years or > 2 years after HDT, ISS stage and standard versus high-risk cytogenetics. The primary end-point of this part of the study is comparison of time to progression in carfilzomib-dexamethasone maintenance arm and in the observational arm. Patients will continue on maintenance therapy/observation until progression, end of study or fulfil standard criteria for discontinuation of treatment according to the protocol.

The study will include 200 patients with relapse of multiple myeloma more than one year after initial HDT. It is a prerequisite that the patients have at least 2.0 x 10m CD34+ stem cells/kg body weight saved in the freezer. The study is conducted by the Nordic Myeloma Study Group (NMSG) at clinics in Denmark, Sweden, Norway, Finland and Lithuania. The first patient was included in January 2015 and enrolment is expected to continue until December 2017. The study ends when the last included patient has been followed for 9 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma diagnosis according to IMWG criteria
* First treatment demanding relapse after HDT according to IMWG criteria
* More than 2.0 x 10m CD34+ stem cells / kg body weight in the freezer for stem cell support
* Signed informed consent given prior to any study related activities have been performed
* Age > 18 years

Exclusion Criteria:

Demographic

* Allogeneic transplantation scheduled as a part of the treatment
* Treatment demanding relapse less than one year after HDT
* Myeloma treatment after the first HDT, except radiotherapy, bisphosphonates, denosumab and corticosteroids less than 6 days for symptom control
* Patients not having received HDT as first line treatment
* Previous treatment with carfilzomib
* Expected survival of less than six months
* Performance status (WHO) ≥ 3

Laboratory

* Serum M-component < 5 g/l and urine M-component < 200 mg/l
* Any of the following laboratory abnormalities:

  * Absolute neutrophil count (ANC) < 1.0 × 109/L
  * Hemoglobin < 5 mmol/L (<80 g/L) (prior RBC transfusion or recombinant human erythropoietin use is permitted)
  * Platelet count < 50 × 109/L (< 30 × 109/L if myeloma involvement in the bone marrow is > 50%)
  * Serum ALT or AST > 3.5 times the upper limit of normal and serum direct bilirubin > 34 µmol/L (2 mg/dL)
  * Creatinine clearance (CrCl) < 15 mL/minute, either measured or calculated using a standard formula

Concurrent conditions

* Concurrent disease making treatment with carfilzomib, cyclophosphamide or dexamethasone unsuitable
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to enrolment
* Major surgery within 21 days prior to enrolment
* Acute active infection requiring treatment
* Known or suspected hypersensitivity or intolerance to melphalan, dexamethasone or Captisol® (a cyclodextrin derivative)
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrolment, NYHA Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, uncontrolled severe arrhythmias, or cardiac amyloidosis
* LVEF <40%, determined by 2-D transthoracic echocardiogram (ECHO) or Multigated Acquisition Scan (MUGA)
* Pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrolment
* Serious hepatic disorder, including active hepatitis B or C infection
* Other serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Use of any investigational agents or experimental medical device within 28 days prior to enrolment into the study

Ethical/other

* Pregnant or lactating females
* Females of childbearing potential must agree to ongoing pregnancy testing and to practice contraception
* Male subjects must agree to practice contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2018-04-23 (Actual); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of time to progression after high-dose melphalan with stem cell support (HDT) performed at diagnosis and time to progression after a salvage HDT combined with carfilzomib-cyclophosphamide-dexamethasone | 3 years
Comparison of time to progression between carfilzomib-dexamethasone maintenance and observation in patients treated with salvage HDT. | 3 years

SECONDARY OUTCOMES:
Adverse events assessed by CTCAE v4.0 in carfilzomib-cyclophosphamide-dexamethasone induction regime and carfilzomib as part of the high-dose melphalan conditioning | 5 months
Response rates of carfilzomib-cyclophosphamide-dexamethasone induction therapy and HDT | 5 months
Time to marrow regeneration (neutrophil- and platelet recovery) after the HDT | 3 weeks
Adverse events assessed by CTCAE v4.0 in maintenance treatment with carfilzomib-dexamethasone | 3 years
Comparison of overall survival between carfilzomib-dexamethasone maintenance and observation in patients treated with a salvage HDT | 3 years
Quality of life assessed by EORTC QLQ-MY20 and EORTC QLQ-C30 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Gregersen, MD, Principal Investigator — Aalborg University Hospital
Locations (5):
- Aalborg University Hospital, Aalborg, Denmark
- Turku University Hospital, Turku, Finland
- Vilnius University hospital "Santariskiu Clinics", Vilnius, Lithuania
- Oslo University Hospital, Oslo, Norway
- Skåne University Hospital, Lund, Sweden